CLINICAL TRIAL: NCT05694884
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial to Evaluate the Efficacy and Safety of Eblasakimab in Male or Female Moderate-to-Severe Atopic Dermatitis Patients Previously Treated With Dupilumab
Brief Title: Study of Eblasakimab in Male or Female Moderate-to-Severe Atopic Dermatitis Patients Previously Treated With Dupilumab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASLAN004-004
Record Dates: First submitted 2023-01-09; First posted 2023-01-23 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; IL-13; ASLAN004; IL-13Rα1; Eczema; Anti-IL-13Rα1; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo loading dose equivalents at Baseline and Week 1, then placebo dose equivalents every week (QW) from Week 2 to Week 15
  Interventions: Drug: Placebo
- ASLAN004 (Experimental): Week 0, 1: LD of 600 mg; Week 2 through Week 15 QW: 400 mg dose
  Interventions: Drug: ASLAN004

INTERVENTIONS:
Drug: Placebo — Placebo Comparator
  Arms: Placebo
Drug: ASLAN004 — ASLAN004
  Arms: ASLAN004

SUMMARY:
Multicenter, randomized, double-blind, placebo-controlled, parallel arm clinical study designed to evaluate the efficacy and safety of eblasakimab in participants with moderate-to-severe atopic dermatitis (AD) previously treated with dupilumab.The study consists of a 16-week treatment period and an 8-week follow-up period up to Week 24. Eligible participants will be randomized into one of the 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 years
* Willing and able to comply with clinic visits and study-related procedures
* Chronic AD present for at least 1 year prior to screening
* Have vIGA score of ≥3 (5-scale of 0 to 4) at baseline
* Have ≥10% BSA of AD involvement at baseline
* Have EASI ≥18 at screening and baseline
* History of inadequate response to, intolerance to or contraindication to a stable regimen of topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) as treatment for AD
* All participants must have previously been treated with dupilumab meeting one of the following conditions:

  1. Participants who stopped dupilumab treatment due to non-response, partial response, loss of efficacy must have been previously treated with dupilumab for at least 16 weeks duration;
  2. Participants who stopped dupilumab treatment due to intolerance or adverse events (AEs) to the drug may enter the study with no required prior length of dupilumab treatment;
  3. Participants who stopped dupilumab treatment due to cost or loss of access to dupilumab or for any other reasons may enter the study with no required prior length of dupilumab treatment;

Exclusion Criteria:

* Use of immunosuppressive/immunomodulating drugs and/or therapies, JAK inhibitors, or phototherapy (including tanning booth/parlor) within 4 weeks prior to the Baseline visit
* Have an uncontrolled chronic disease that may require multiple intermittent use of systemic corticosteroids at Screening, as defined by the Investigator
* Have uncontrolled asthma that might require bursts of oral or systemic corticosteroids, or require either of the following due to ≥1 exacerbations within 12 months before Baseline:

  1. Systemic (oral and/or parenteral) corticosteroid treatment;
  2. Hospitalization for >24 hours;
* Have had systemic treatment with small molecule investigational drugs within 8 weeks or 5 half-lives (if known), whichever is longer, prior to the Baseline visit
* Have received treatment with topical corticosteroids (TCS), topical calcineurin inhibitors (TCI) such as tacrolimus and pimecrolimus, topical phosphodiesterase inhibitors such as crisaborole, topical JAK inhibitors (commercial or investigational use), within 1 week prior to randomization
* Have inadequate organ function or abnormal lab results considered clinically significant by the Investigator at the Screening visit
* History of human immunodeficiency virus (HIV) or positive HIV serology at Screening
* Infected with hepatitis B or hepatitis C viruses. For Hepatitis B, all subjects will undergo testing for Hepatitis B Surface Antigen (HBsAg) and Hepatitis B Core Antibody (HBcAb) during Screening. Subjects who are HBsAg positive are not eligible for the study. Subjects who are HBsAg negative and HBcAb positive will be tested for Hepatitis B Surface Antibody (HBsAb) and if HBsAb is positive, may be enrolled in the study; if HBsAb is negative, the subject is not eligible for the study. For Hepatitis C, all subjects will undergo testing for Hepatitis C antibody (HCVAb) during Screening. Subjects who are HCVAb positive are not eligible for the study. Active COVID-19 infection at Baseline.
* Have known liver cirrhosis and/or chronic hepatitis of any etiology
* Known diagnosis of active tuberculosis or non-tuberculous mycobacterial infection or latent tuberculosis unless it is well documented by a specialist that the patient has been adequately treated
* Allergen immunotherapy should be discontinued 6 months before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Percent change from Baseline in Eczema Area and Severity Index (EASI) at Week 16 | Baseline, Week 16
  The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD

SECONDARY OUTCOMES:
Proportion of participants achieving validated Investigator's Global Assessment (vIGA) response of 0 (clear) or 1 (almost clear) at Week 16 | Week 16
  IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear)
Proportion of participants with a 75% reduction Eczema Area and Severity Index 75 (EASI) | Week 16
  EASI scores range from 0 to 72 (severe)The EASI responder is defined as a participant who achieves a ≥75% improvement (EASI 75) from baseline in the EASI score
Proportion of participants achieving EASI 50 | Week 16
  EASI scores range from 0 to 72 (severe)The EASI responder is defined as a participant who achieves a ≥50% improvement (EASI 50) from baseline in the EASI score
Proportion of participants achieving EASI 90 | Week 16
  EASI scores range from 0 to 72 (severe)The EASI responder is defined as a participant who achieves a ≥90% improvement (EASI 90) from baseline in the EASI score
Proportion of participants with EASI <7 | Week 16
  EASI scores range from 0 to 72 (severe)
Absolute and percent change in peak Pruritus Numerical Rating Scale (P-NRS) | Week 16 and Week 24
  The P-NRS is an 11-point scale used by patients to assess their worst itch severity over the past 24 hours, with 0 indicating no itch and 10 indicating the worst itch imaginable. Pruritus assessments will be recorded daily by the patient using an electronic diary
Proportion of participants achieving a 4-point reduction in peak Pruritus Numerical Rating Scale | Week 16
  Pruritus Numerical Rating Scale
Change in Body Surface Area (BSA) affected with AD | Week 16 and Week 24
  BSA ranges from 0% to 100 % with higher values representing greater extent of AD
Change in SCORing Atopic Dermatitis (SCORAD) | Week 16 and Week 24
  The SCORAD is a validated measure of the extent and severity of atopic dermatitis lesions, along with subjective symptoms. The score ranges from 0 to 103, with higher values indicating a more extensive and/or severe condition
Change in Dermatology Life Quality Index (DLQI) | Week 16 and Week 24
  The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the patient's perception of the impact of AD disease symptoms and treatment on their quality of life (QoL). The 10 questions assess QoL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease). A high score is indicative of a poor QoL
Change in Patient-Oriented Eczema Measure (POEM) | Week 16 and Week 24
  The POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor QoL)
Change in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Index Score United States and United Kingdom Algorithm | Week 16 and Week 24
  The EQ-5D-5L is a 2-part measurement. The second part is assessed using a visual analog scale (VAS) that ranges from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine
Absolute and percent change in sleep disturbance numerical rating scale (SD-NRS) | Week 16 and Week 24
  The SD-NRS is an 11-point scale used by patients to assess their sleep disturbance severity over the past 24 hours, with 0 indicating no or minimal sleep disturbance and 10 indicating the worst imaginable sleep disturbance. SD-NRS assessments will be recorded daily by the patient using an electronic diary
Proportion of participants achieving a 4-point reduction in sleep disturbance numerical rating scale | Week 16
Percent change from baseline of validated Investigator's Global Assessment (vIGA) | Week 24
  IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear)
Percent change from baseline of Eczema Area and Severity Index | Week 24
  EASI scores range from 0 to 72 (severe)
Number of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) from study drug administration | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — ASLAN Pharmaceuticals
Locations (26):
- United States (23):
  - ASLAN Investigative Site, Birmingham, Alabama
  - ASLAN Investigative Site, Encino, California
  - ASLAN Investigative Site, Fountain Valley, California
  - ASLAN Investigative Site, Long Beach, California
  - ASLAN Investigative Site, Los Angeles, California
  - ASLAN Investigative Site, Sherman Oaks, California
  - ASLAN Investigative Site, Boca Raton, Florida
  - ASLAN Investigative Site, Hollywood, Florida
  - ASLAN Investigative Site, Miami Lakes, Florida
  - ASLAN Investigative Site, North Miami Beach, Florida
  - ASLAN Investigative Site, Orange City, Florida
  - ASLAN Investigative Site, Saint Augustine, Florida
  - ASLAN Investigative Site, St. Petersburg, Florida
  - ASLAN Investigative Site, New Albany, Indiana
  - ASLAN Investigative Site, Louisville, Kentucky
  - ASLAN Investigative Site, Quincy, Massachusetts
  - ASLAN Investigative Site, Auburn Hills, Michigan
  - ASLAN Investigative Site, Las Vegas, Nevada
  - ASLAN Investigative Site, East Amherst, New York
  - ASLAN Investigative Site, Charlotte, North Carolina
  - ASLAN Investigative Site, Oklahoma City, Oklahoma
  - ASLAN Investigative Site, Johnston, Rhode Island
  - ASLAN Investigative Site, Charleston, South Carolina
- Canada (3):
  - ASLAN Investigative Site, Hamilton, Ontario
  - ASLAN Investigative Site, Ottawa, Ontario
  - ASLAN Investigative Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No